CLINICAL TRIAL: NCT01159769
Title: Patient Perceptions and Quality of Life Associated With the Use of Olapatadine 0.2% for the Treatment of Allergic Conjunctivitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SMA-10-13
Record Dates: First submitted 2010-07-08; First posted 2010-07-09 (Estimated); Results first posted 2012-04-03 (Estimated); Last update posted 2012-04-03 (Estimated); Status verified 2012-03

CONDITIONS: Allergic Conjunctivitis
Keywords: Allergic conjunctivitis
MeSH Terms: conditions — Conjunctivitis, Allergic | interventions — Olopatadine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Olopatadine 0.2% (Experimental): 1 drop self-administered in each eye once daily in the morning for 7 days
  Interventions: Drug: Olopatadine hydrochloride ophthalmic solution, 0.2% (Pataday®)

INTERVENTIONS:
Drug: Olopatadine hydrochloride ophthalmic solution, 0.2% (Pataday®) — Commercially marketed ophthalmic solution for the treatment of ocular itching associated with allergic conjunctivitis
  Other Names: Pataday®

SUMMARY:
The purpose of this study is to evaluate patient perceptions of olopatadine 0.2% dosed once daily in patients previously treated with twice-daily, topical, ocular, anti-allergy medications.

ELIGIBILITY:
Inclusion Criteria:

* 12 years of age or older.
* History (within the past 24 months) of allergic conjunctivitis.
* Active signs and symptoms of ocular allergies.
* Ocular health within normal limits, as determined by the investigator or subinvestigator.
* Willing to avoid contact lens wear each study visit immediately prior to study medication instillation and for 10 minutes after instillation of study drug.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Contraindications or hypersensitivity to study medication or its components.
* One sighted eye or not correctable to 0.6 logMAR or better in both eyes at the screening visit.
* Known history of recurrent corneal erosion syndrome.
* Ocular trauma or surgical intervention within 6 months prior to Visit 1.
* Participation in any other investigational study within 30 days before Visit 1.
* Pregnant or nursing.
* Other protocol-defined exclusion criteria may apply.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2010-06; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from 12 US study centers. Eligible patients having a history of allergic conjunctivitis and treated with protocol-specified anti-allergy medications for at least 7 days within 6 months prior to Visit 1 were enrolled. Investigators reviewed files to identify patients.
Pre-assignment Details: 215 patients were enrolled. All patients received the same treatment.
Period: Overall Study
Arm/Group | Olopatadine 0.2%
Started | 215
Completed | 214
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Olopatadine 0.2%
Number analyzed (Participants) | 215
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7
  Between 18 and 65 years | 127
  >=65 years | 81
Age Continuous [Mean (Standard Deviation); unit: years] | 55.03 (18.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 141
  Male | 74

OUTCOME MEASURES:

1. Primary Outcome: Overall Patient Satisfaction
Description: Overall satisfaction was assessed by the patient on a questionnaire. The patient was instructed to select a single response to the statement, "Overall, how satisfied are you with your current eye allergy medication?" A 5-point scale was used: very satisfied, satisfied, undecided, dissatisfied, very dissatisfied. Results are reported as the percentage of patients who responded, "very satisfied" or "satisfied."
Time Frame: Day 0
Population: All subjects who used the study medication at least once (intent to treat).
Measure: Number; unit: Percentage of Participants
Arm/Group | Olopatadine 0.2%
Number analyzed (Participants) | 214
Percentage of Participants | 70.1

2. Primary Outcome: Overall Patient Satisfaction
Description: Overall satisfaction was assessed by the patient on a questionnaire. The patient was instructed to select a single response to the statement, "Overall, how satisfied were you with olopatadine 0.2%?" A 5-point scale was used: very satisfied, satisfied, undecided, dissatisfied, very dissatisfied. Results are reported as the percentage of patients who responded, "very satisfied" or "satisfied."
Time Frame: Day 7
Population: All subjects who used the study medication at least once (intent to treat).
Measure: Number; unit: Percentage of Participants
Arm/Group | Olopatadine 0.2%
Number analyzed (Participants) | 214
Percentage of Participants | 89.3

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the study: 7 June 2010 to 7 August 2010.
Description: This reporting group includes all subjects who used the study medication at least once (intent to treat). Subjects were queried about any symptoms that would suggest an adverse event with, "Have you had any health problems since your last study visit?" and "Have there been any changes in the medicines you take since your last study visit?"
Arm/Group | Olopatadine 0.2%
Serious Adverse Events (participants affected / at risk) | 2/215
Other Adverse Events (participants affected / at risk) | 0/215
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Olopatadine 0.2% (N=215)
Stomach pain (Gastrointestinal disorders) | 1 — Unrelated
Colorectal cancer (Gastrointestinal disorders) | 1 — Unrelated

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Alcon reserves the right of prior review of any publication or presentation of information related to the study.